CLINICAL TRIAL: NCT04461184
Title: The Great Plains Internet Wellness Study for Aging: The GP I-WAS Project
Brief Title: The Great Plains Internet Wellness Study for Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Principal Investigator, Ryan McGrath, Assistant Professor, North Dakota State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NorthDakotaSU
Record Dates: First submitted 2020-06-25; First posted 2020-07-08 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Internet Based Wellness Program; Obesity; Adult Population
MeSH Terms: conditions — Obesity | interventions — Aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet wellness intervention for aging (Experimental): Feasibility components will be evaluated with a 5-point Likert scale may include open ended items for more detailed feedback. Participants will be asked to visit NDSU at the beginning and end of the intervention, and at 1-month follow-up. After written informed consent, each participant will complete a descriptive questionnaire at the beginning of the intervention period, and a health-related questionnaire at the beginning and end of the intervention, and at follow-up that includes self-rated health, current smoking status, smoking history, alcohol use, morbid conditions, functional disability, and depression status. Standing height and waist circumference will be collected with a tape measure. Body weight and composition will be measured with the InBody 570. Anthropometric and body composition assessments will be collected pre, post, and follow up.
  Interventions: Behavioral: Internet Wellness Intervention for Aging

INTERVENTIONS:
Behavioral: Internet Wellness Intervention for Aging — Internet technologies have emerged as a platform for performing wellness interventions that also have wide outreach. Previous studies that have used the internet for delivering health interventions have found that older adults valued this platform, used it for researching health information and social communications. Likewise, the effectiveness of delivering health-related information intended for behavior change through the internet is equal to that of print-based delivery, thereby lowering costs and expanding reach. Thus, the internet provides a unique platform for conducting interventions. The internet based wellness intervention will be a low cost method focused on older adults to help increase intrinsic motivation through autonomy, competence, and relatedness (Intrinsic Motivation) to help increase daily physical activity.

SUMMARY:
Obesity is a major public health concern in older adults, who are also one of the fastest growing populations in the United States. Engaging in healthy behaviors such as physical activity, a healthy diet, and adequate sleep have each shown to be influential in reducing obesity. The internet could be an effective tool for administering a wellness intervention for older adults. Our goal is to help older adults achieve healthy lifestyles that promote successful aging.

DETAILED DESCRIPTION:
Obesity is a major public health concern in older adults, who are also one of the fastest growing populations in the United States. The health consequences associated with obesity in older adulthood are severe and include increased risk for chronic diseases, poor physical functioning and early mortality. Concurrently engaging in healthy behaviors such as physical activity, a healthy diet, and adequate sleep have each shown to be influential in reducing obesity. Despite evidence suggesting that these healthy behaviors reduce the risk for obesity, older adults have difficulty achieving such healthy lifestyles due to barriers such as geographical isolation from lack of transportation, motivation and education. The internet is an effective mode for relaying health information to a wide-ranging audience, including those that live in rural communities or are home bound. Further, internet usage among older adults continues to increase. Therefore, the internet could be an effective tool for administering a wellness intervention for older adults and incorporating community-based participatory research principles such as inviting stakeholders (i.e., older adults) in all phases of the research will magnify the impact of the research for the population in which it is intended to help. Our long-term goal is to help older adults achieve healthy lifestyles that promote successful aging. The overall objective of the proposed research, which is the next step in pursuit of that goal, is to improve healthy lifestyles in older adults by utilizing the internet for delivering a wellness intervention that is designed by both investigators and stakeholders. To propel toward accomplishing our overall objective, the following three specific aims will be pursued: 1) collaborate with stakeholders in all phases of the internet-based wellness intervention to gain knowledge on the perspectives of the older adult population, 2) assess the feasibility of an internet-based wellness intervention for obese older adults, and 3) determine if completing an internet based wellness intervention improves healthy behaviors among obese older adults. We will recruit 20 eligible older adults to participate in an internet-based wellness intervention. A prospective, within-participant design with multiple assessments across the 10-week study period and 1-month follow-up will allow us to optimize power with a smaller sample size and assess within-person change over time.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged at least 65 years that can use the internet daily, have a body mass index of ≥ 30 kg/m2, and are apparently healthy (i.e., medically able to participate in physical activity as determined by the PAR-Q+) Will be eligible for the study.

Exclusion Criteria:

* Those with a surgical implant, who are unable to read or speak the English language fluently, with a severe cognitive impairment, and unable to wear an accelerometer on their waist will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Increase Physical Activity and Participation | 10-weeks
  Actigraph accelerometer and physical activity recall will be used to measure and record physical activity throughout the 10-week internet wellness intervention.
Create a more balanced dietary intake based on nutrient dense foods | 10-weeks
  Participants will complete the Arizona Food Frequency Questionnaire (AFFQ) to assess dietary intake at the beginning and end of the intervention, and at 1-month follow-up. The AFFQ is a modified version of the Health Habits Questionnaire and has demonstrated strong reliability and validity for assessing dietary intake. In addition, each report will contain a personalized message from the dietitian to each participant. Intake of nutritionally dense foods (e.g., vegetables, lean proteins) and decreased intake of calorically dense foods (e.g., high sugar foods) will be compared to assess dietary change.

CONTACTS AND LOCATIONS:
Locations (1):
- North Dakota State University Health, Nutrition, and Exercise Sciences, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill JO, Catenacci V, Wyatt HR. Obesity: overview of an epidemic. Psychiatr Clin North Am. 2005 Mar;28(1):1-23, vii. doi: 10.1016/j.psc.2004.09.010. No abstract available. PMID 15733608
- [Background] Fakhouri TH, Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity among older adults in the United States, 2007-2010. NCHS Data Brief. 2012 Sep;(106):1-8. PMID 23102091
- [Background] Zamboni M, Mazzali G, Fantin F, Rossi A, Di Francesco V. Sarcopenic obesity: a new category of obesity in the elderly. Nutr Metab Cardiovasc Dis. 2008 Jun;18(5):388-95. doi: 10.1016/j.numecd.2007.10.002. Epub 2008 Apr 18. PMID 18395429
- [Background] Saint Onge JM, Krueger PM. Health Lifestyle Behaviors among U.S. Adults. SSM Popul Health. 2017 Dec;3:89-98. doi: 10.1016/j.ssmph.2016.12.009. PMID 28785602
- [Background] Hargens TA, Kaleth AS, Edwards ES, Butner KL. Association between sleep disorders, obesity, and exercise: a review. Nat Sci Sleep. 2013 Mar 1;5:27-35. doi: 10.2147/NSS.S34838. Print 2013. PMID 23620691
- [Background] Bales CW, Porter Starr KN. Obesity Interventions for Older Adults: Diet as a Determinant of Physical Function. Adv Nutr. 2018 Mar 1;9(2):151-159. doi: 10.1093/advances/nmx016. PMID 29659687
- [Background] Batsis JA, Zagaria AB. Addressing Obesity in Aging Patients. Med Clin North Am. 2018 Jan;102(1):65-85. doi: 10.1016/j.mcna.2017.08.007. Epub 2017 Oct 21. PMID 29156188
- [Background] Cohen SA, Greaney ML, Sabik NJ. Assessment of dietary patterns, physical activity and obesity from a national survey: Rural-urban health disparities in older adults. PLoS One. 2018 Dec 5;13(12):e0208268. doi: 10.1371/journal.pone.0208268. eCollection 2018. PMID 30517166
- [Background] Douthit N, Kiv S, Dwolatzky T, Biswas S. Exposing some important barriers to health care access in the rural USA. Public Health. 2015 Jun;129(6):611-20. doi: 10.1016/j.puhe.2015.04.001. Epub 2015 May 27. PMID 26025176
- [Background] Befort CA, Nazir N, Perri MG. Prevalence of obesity among adults from rural and urban areas of the United States: findings from NHANES (2005-2008). J Rural Health. 2012 Fall;28(4):392-7. doi: 10.1111/j.1748-0361.2012.00411.x. Epub 2012 May 31. PMID 23083085
- [Background] Bolin JN, Bellamy GR, Ferdinand AO, Vuong AM, Kash BA, Schulze A, Helduser JW. Rural Healthy People 2020: New Decade, Same Challenges. J Rural Health. 2015 Summer;31(3):326-33. doi: 10.1111/jrh.12116. Epub 2015 May 7. PMID 25953431
- [Background] Jones RB, Ashurst EJ, Atkey J, Duffy B. Older people going online: its value and before-after evaluation of volunteer support. J Med Internet Res. 2015 May 18;17(5):e122. doi: 10.2196/jmir.3943. PMID 25986724
- [Background] Marcus BH, Lewis BA, Williams DM, Dunsiger S, Jakicic JM, Whiteley JA, Albrecht AE, Napolitano MA, Bock BC, Tate DF, Sciamanna CN, Parisi AF. A comparison of Internet and print-based physical activity interventions. Arch Intern Med. 2007 May 14;167(9):944-9. doi: 10.1001/archinte.167.9.944. PMID 17502536
- [Background] Jonkman NH, van Schooten KS, Maier AB, Pijnappels M. eHealth interventions to promote objectively measured physical activity in community-dwelling older people. Maturitas. 2018 Jul;113:32-39. doi: 10.1016/j.maturitas.2018.04.010. Epub 2018 Apr 25. PMID 29903646
- [Background] Rogers MA, Lemmen K, Kramer R, Mann J, Chopra V. Internet-Delivered Health Interventions That Work: Systematic Review of Meta-Analyses and Evaluation of Website Availability. J Med Internet Res. 2017 Mar 24;19(3):e90. doi: 10.2196/jmir.7111. PMID 28341617
- [Background] Schoeppe S, Alley S, Van Lippevelde W, Bray NA, Williams SL, Duncan MJ, Vandelanotte C. Efficacy of interventions that use apps to improve diet, physical activity and sedentary behaviour: a systematic review. Int J Behav Nutr Phys Act. 2016 Dec 7;13(1):127. doi: 10.1186/s12966-016-0454-y. PMID 27927218
- [Background] Pontzer H, Durazo-Arvizu R, Dugas LR, Plange-Rhule J, Bovet P, Forrester TE, Lambert EV, Cooper RS, Schoeller DA, Luke A. Constrained Total Energy Expenditure and Metabolic Adaptation to Physical Activity in Adult Humans. Curr Biol. 2016 Feb 8;26(3):410-7. doi: 10.1016/j.cub.2015.12.046. Epub 2016 Jan 28. PMID 26832439
- [Background] Jakicic JM, Rogers RJ, Davis KK, Collins KA. Role of Physical Activity and Exercise in Treating Patients with Overweight and Obesity. Clin Chem. 2018 Jan;64(1):99-107. doi: 10.1373/clinchem.2017.272443. Epub 2017 Nov 20. PMID 29158251
- [Background] Wiklund P. The role of physical activity and exercise in obesity and weight management: Time for critical appraisal. J Sport Health Sci. 2016 Jun;5(2):151-154. doi: 10.1016/j.jshs.2016.04.001. Epub 2016 Apr 8. PMID 30356545
- [Background] Ness-Abramof R, Apovian CM. Diet modification for treatment and prevention of obesity. Endocrine. 2006 Feb;29(1):5-9. doi: 10.1385/endo:29:1:5. PMID 16622287
- [Background] Beccuti G, Pannain S. Sleep and obesity. Curr Opin Clin Nutr Metab Care. 2011 Jul;14(4):402-12. doi: 10.1097/MCO.0b013e3283479109. PMID 21659802
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Horowitz CR, Robinson M, Seifer S. Community-based participatory research from the margin to the mainstream: are researchers prepared? Circulation. 2009 May 19;119(19):2633-42. doi: 10.1161/CIRCULATIONAHA.107.729863. PMID 19451365
- [Background] Ryan K, Dockray S, Linehan C. A systematic review of tailored eHealth interventions for weight loss. Digit Health. 2019 Feb 5;5:2055207619826685. doi: 10.1177/2055207619826685. eCollection 2019 Jan-Dec. PMID 30783535
- [Background] Ghanvatkar S, Kankanhalli A, Rajan V. User Models for Personalized Physical Activity Interventions: Scoping Review. JMIR Mhealth Uhealth. 2019 Jan 16;7(1):e11098. doi: 10.2196/11098. PMID 30664474
- [Background] Gardner B, Lally P, Wardle J. Making health habitual: the psychology of 'habit-formation' and general practice. Br J Gen Pract. 2012 Dec;62(605):664-6. doi: 10.3399/bjgp12X659466. No abstract available. PMID 23211256
- [Background] Riffin C, Kenien C, Ghesquiere A, Dorime A, Villanueva C, Gardner D, Callahan J, Capezuti E, Reid MC. Community-based participatory research: understanding a promising approach to addressing knowledge gaps in palliative care. Ann Palliat Med. 2016 Jul;5(3):218-24. doi: 10.21037/apm.2016.05.03. PMID 27481321
- [Background] Wallerstein NB, Duran B. Using community-based participatory research to address health disparities. Health Promot Pract. 2006 Jul;7(3):312-23. doi: 10.1177/1524839906289376. Epub 2006 Jun 7. PMID 16760238
- [Background] Salimi Y, Shahandeh K, Malekafzali H, Loori N, Kheiltash A, Jamshidi E, Frouzan AS, Majdzadeh R. Is Community-based Participatory Research (CBPR) Useful? A Systematic Review on Papers in a Decade. Int J Prev Med. 2012 Jun;3(6):386-93. PMID 22783464
- [Background] Hernandez DC, Johnston CA. Individual and Environmental Barriers to Successful Aging: The Importance of Considering Environmental Supports. Am J Lifestyle Med. 2016 Oct 24;11(1):21-23. doi: 10.1177/1559827616672617. eCollection 2017 Jan-Feb. PMID 30202307
- [Background] Bennett JA, Winters-Stone K. Motivating older adults to exercise: what works? Age Ageing. 2011 Mar;40(2):148-9. doi: 10.1093/ageing/afq182. Epub 2011 Jan 20. No abstract available. PMID 21252038
- [Background] Nicklett EJ, Kadell AR. Fruit and vegetable intake among older adults: a scoping review. Maturitas. 2013 Aug;75(4):305-12. doi: 10.1016/j.maturitas.2013.05.005. Epub 2013 Jun 12. PMID 23769545
- [Background] Sheeran P, Maki A, Montanaro E, Avishai-Yitshak A, Bryan A, Klein WM, Miles E, Rothman AJ. The impact of changing attitudes, norms, and self-efficacy on health-related intentions and behavior: A meta-analysis. Health Psychol. 2016 Nov;35(11):1178-1188. doi: 10.1037/hea0000387. Epub 2016 Jun 9. PMID 27280365
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Teixeira PJ, Carraca EV, Markland D, Silva MN, Ryan RM. Exercise, physical activity, and self-determination theory: a systematic review. Int J Behav Nutr Phys Act. 2012 Jun 22;9:78. doi: 10.1186/1479-5868-9-78. PMID 22726453
- [Background] Teixeira PJ, Silva MN, Mata J, Palmeira AL, Markland D. Motivation, self-determination, and long-term weight control. Int J Behav Nutr Phys Act. 2012 Mar 2;9:22. doi: 10.1186/1479-5868-9-22. PMID 22385818
- [Background] Jopp DS, Jung S, Damarin AK, Mirpuri S, Spini D. Who Is Your Successful Aging Role Model? J Gerontol B Psychol Sci Soc Sci. 2017 Mar 1;72(2):237-247. doi: 10.1093/geronb/gbw138. PMID 27803026
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Ling CH, de Craen AJ, Slagboom PE, Gunn DA, Stokkel MP, Westendorp RG, Maier AB. Accuracy of direct segmental multi-frequency bioimpedance analysis in the assessment of total body and segmental body composition in middle-aged adult population. Clin Nutr. 2011 Oct;30(5):610-5. doi: 10.1016/j.clnu.2011.04.001. Epub 2011 May 8. PMID 21555168
- [Background] Sartorio A, Malavolti M, Agosti F, Marinone PG, Caiti O, Battistini N, Bedogni G. Body water distribution in severe obesity and its assessment from eight-polar bioelectrical impedance analysis. Eur J Clin Nutr. 2005 Feb;59(2):155-60. doi: 10.1038/sj.ejcn.1602049. PMID 15340370
- [Background] Montoye AHK, Nelson MB, Bock JM, Imboden MT, Kaminsky LA, Mackintosh KA, McNarry MA, Pfeiffer KA. Raw and Count Data Comparability of Hip-Worn ActiGraph GT3X+ and Link Accelerometers. Med Sci Sports Exerc. 2018 May;50(5):1103-1112. doi: 10.1249/MSS.0000000000001534. PMID 29283934
- [Background] Tudor-Locke C, Camhi SM, Troiano RP. A catalog of rules, variables, and definitions applied to accelerometer data in the National Health and Nutrition Examination Survey, 2003-2006. Prev Chronic Dis. 2012;9:E113. doi: 10.5888/pcd9.110332. Epub 2012 Jun 14. PMID 22698174
- [Background] Choi L, Liu Z, Matthews CE, Buchowski MS. Validation of accelerometer wear and nonwear time classification algorithm. Med Sci Sports Exerc. 2011 Feb;43(2):357-64. doi: 10.1249/MSS.0b013e3181ed61a3. PMID 20581716
- [Background] Sasaki JE, John D, Freedson PS. Validation and comparison of ActiGraph activity monitors. J Sci Med Sport. 2011 Sep;14(5):411-6. doi: 10.1016/j.jsams.2011.04.003. Epub 2011 May 25. PMID 21616714
- [Background] Kozey-Keadle S, Libertine A, Lyden K, Staudenmayer J, Freedson PS. Validation of wearable monitors for assessing sedentary behavior. Med Sci Sports Exerc. 2011 Aug;43(8):1561-7. doi: 10.1249/MSS.0b013e31820ce174. PMID 21233777
- [Background] Rosenberger ME, Buman MP, Haskell WL, McConnell MV, Carstensen LL. Twenty-four Hours of Sleep, Sedentary Behavior, and Physical Activity with Nine Wearable Devices. Med Sci Sports Exerc. 2016 Mar;48(3):457-65. doi: 10.1249/MSS.0000000000000778. PMID 26484953
- [Background] Keadle SK, Shiroma EJ, Freedson PS, Lee IM. Impact of accelerometer data processing decisions on the sample size, wear time and physical activity level of a large cohort study. BMC Public Health. 2014 Nov 24;14:1210. doi: 10.1186/1471-2458-14-1210. PMID 25421941
- [Background] Cole RJ, Kripke DF, Gruen W, Mullaney DJ, Gillin JC. Automatic sleep/wake identification from wrist activity. Sleep. 1992 Oct;15(5):461-9. doi: 10.1093/sleep/15.5.461. PMID 1455130
- [Background] Ainsworth BE, Haskell WL, Whitt MC, Irwin ML, Swartz AM, Strath SJ, O'Brien WL, Bassett DR Jr, Schmitz KH, Emplaincourt PO, Jacobs DR Jr, Leon AS. Compendium of physical activities: an update of activity codes and MET intensities. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S498-504. doi: 10.1097/00005768-200009001-00009. PMID 10993420
- [Background] Gomersall SR, Olds TS, Ridley K. Development and evaluation of an adult use-of-time instrument with an energy expenditure focus. J Sci Med Sport. 2011 Mar;14(2):143-8. doi: 10.1016/j.jsams.2010.08.006. Epub 2010 Oct 6. PMID 20932797
- [Background] Mace CJ, Maddison R, Olds T, Kerse N. Validation of a computerized use of time recall for activity measurement in advanced-aged adults. J Aging Phys Act. 2014 Apr;22(2):245-54. doi: 10.1123/japa.2012-0280. Epub 2013 May 22. PMID 23752221
- [Background] Foley LS, Maddison R, Rush E, Olds TS, Ridley K, Jiang Y. Doubly labeled water validation of a computerized use-of-time recall in active young people. Metabolism. 2013 Jan;62(1):163-9. doi: 10.1016/j.metabol.2012.07.021. Epub 2012 Sep 11. PMID 22980224
- [Background] Thomson CA, Giuliano A, Rock CL, Ritenbaugh CK, Flatt SW, Faerber S, Newman V, Caan B, Graver E, Hartz V, Whitacre R, Parker F, Pierce JP, Marshall JR. Measuring dietary change in a diet intervention trial: comparing food frequency questionnaire and dietary recalls. Am J Epidemiol. 2003 Apr 15;157(8):754-62. doi: 10.1093/aje/kwg025. PMID 12697580
- [Background] Block G, Hartman AM, Dresser CM, Carroll MD, Gannon J, Gardner L. A data-based approach to diet questionnaire design and testing. Am J Epidemiol. 1986 Sep;124(3):453-69. doi: 10.1093/oxfordjournals.aje.a114416. PMID 3740045
- See also: Projections of the Size and Composition of the US Population: 2014 to 2060 — https://mronline.org/wp-content/uploads/2019/08/p25-1143.pdf
- See also: Obesity in Elderly — https://www.ncbi.nlm.nih.gov/sites/books/NBK532533/
- See also: Obesity in older adults — http://citeseerx.ist.psu.edu/viewdoc/download?doi=10.1.1.738.2737&rep=rep1&type=pdf
- See also: Web-based physical activity interventions for older adults: A review. — http://doras.dcu.ie/20896/1/Wani-paper.pdf
- See also: Statistical power analysis for the behavioral sciences. — http://lab.rockefeller.edu/cohenje/PDFs/159CohenBigFishLittleFishTheSciences1989.pdf
- See also: Self-determination theory: A macrotheory of human motivation, development, and health. — http://citeseerx.ist.psu.edu/viewdoc/download?doi=10.1.1.996.3690&rep=rep1&type=pdf
- See also: United States Department of Health and Human Services — https://www.usability.gov/
- See also: l. Assessing sleep using hip and wrist actigraphy — https://link.springer.com/content/pdf/10.1111/sbr.12103.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT04461184/Prot_SAP_000.pdf